CLINICAL TRIAL: NCT00610584
Title: Acupuncture for Seasonal Allergic Rhinitis (ACUSAR) - A Randomised Controlled Trial
Brief Title: Acupuncture for Seasonal Allergic Rhinitis
Acronym: ACUSAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Benno Brinkhaus, Prof. MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EA1/214/07; DFG
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: seasonal allergic rhinitis; acupuncture; RCT; CAM
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Acupuncture Therapy; Cetirizine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): verum acupuncture plus rescue medication (up to 2 doses of second-generation oral antihistamines daily (e.g. 2 x 1 cetirizine dihydrochloride/daily))
  Interventions: Procedure: acupuncture
- 2 (Placebo Comparator): minimal (sham) acupuncture plus rescue medication (up to 2 doses of second-generation oral antihistamines daily (e.g. 2 x 1 cetirizine dihydrochloride/daily))
  Interventions: Procedure: minimal (sham)acupuncture
- 3 (Active Comparator): rescue medication (up to 2 doses of second-generation oral antihistamines daily (e.g. 2 x 1 cetirizine dihydrochloride/daily))alone
  Interventions: Drug: cetirizine dihydrochloride (rescue medication)

INTERVENTIONS:
Procedure: acupuncture — arm 1: verum acupuncture group: 12 interventions (semi-standardised): 8 in the first 4 weeks and 4 in the next 4 weeks + rescue medication (up to 2 doses of second-generation oral antihistamines daily (e.g. 2 x 1 cetirizine dihydrochloride/daily))
  Arms: 1
Procedure: minimal (sham)acupuncture — arm 2: minimal (sham) acupuncture group: 12 interventions (standardised): 8 in the first 4 weeks and 4 in the next 4 weeks + rescue medication (up to 2 doses of second-generation oral antihistamines daily (e.g. 2 x 1 cetirizine dihydrochloride/daily))
  Arms: 2
Drug: cetirizine dihydrochloride (rescue medication) — arm 3: rescue medication (up to 2 doses of second-generation oral antihistamines daily (e.g. 2 x 1 cetirizine dihydrochloride/daily)) alone
  Arms: 3

SUMMARY:
Acupuncture is widely use by patients with seasonal allergic rhinitis (SAR), although there is only limited evidence of its effectiveness. The aim of this three armed randomised controlled multicentre trial is to investigate the efficacy of acupuncture plus rescue medication vs. minimal (sham) acupuncture plus rescue medication vs. (b) rescue medication alone in the treatment of seasonal allergic rhinitis.

DETAILED DESCRIPTION:
Acupuncture is widely use by patients with seasonal allergic rhinitis (SAR), although there is only limited evidence of its effectiveness. The aims of this 3-armed, randomised controlled trial are to investigate whether acupuncture plus rescue medication is non-inferior (closed testing procedure: in case of success in non-inferiority: test of superiority) to minimal acupuncture plus rescue medication in the treatment of SAR (closed testing procedure: closed testing procedure: in case of success in non-inferiority: test of superiority), and whether acupuncture plus rescue medication is non-inferior to rescue medication alone consisting only of oral antihistamines for this indication. The trial interventions will be performed in approximately 40 outpatient centres in Germany. In total, 400 patients with SAR will be randomised to one of three groups: acupuncture plus rescue medication, minimal acupuncture (i.e. superficial needling at non-acupuncture points) plus rescue medication, or rescue medication only. Rescue medication will consist of oral antihistamines. Acupuncture and minimal acupuncture will be administered by physicians specialised in acupuncture and will consist of 12 sessions per patient in the first 8 weeks. Patients in the rescue medication group will receive 12 sessions of acupuncture after 8 weeks. The primary outcome measures will be the mean of Rhinitis Quality of Life Questionnaire score (RQLQ scores between weeks 6 and 8 of the first year (adjusted for baseline values) and the Rescue Medication Score (RMS) between weeks 6 and 8 of the first year (adjusted for baseline values).

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients (aged 16-45 years) with seasonal allergic rhinitis, clinically positive and test positive (skin-prick test and/or RAST) to grass and birch pollen
* Patients with >2 years of moderate to severe SAR
* Positive skin-prick test and/or RAST (at least class 2) results
* Visual analogue scale >40mm and <80 mm for SAR symptoms during the past year
* Patients must be able to complete a diary for self-evaluation of symptoms and recording use of anti-symptomatic medication
* Use of, or indication for, oral antihistamines as anti-allergic medication
* Written informed consent

Exclusion Criteria:

* Perennial SAR or other types of chronic rhinitis
* Allergic asthma and/or moderate to severe atopic dermatitis
* Active tuberculosis
* Autoimmune disorders
* Severe chronic inflammatory diseases
* History of anaphylactic reactions
* Hypersensitivity to Rescue medication or related drugs used in study related drugs
* Specific immunotherapy >3 years
* Simultaneous participation in other clinical trials
* Serious acute or chronic organic disease or mental disorder
* Pregnancy or breast feeding
* Allergy desensitisation therapy (current, during the past two years, or planned in the next two years)
* Blood coagulation disorder and/or current use of anticoagulants
* Previous acupuncture treatment for SAR
* Any Complementary and alternative medicine treatment at the moment, in the last three months or planned in the next two years

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 422 (Actual)
Dates: Start 2008-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Rhinitis Quality of Life Questionnaire score (RQLQ scores between weeks 6 and 8 of the first year (adjusted for baseline values) and the Rescue Medication Score between weeks 6 and 8 of the first year (adjusted for baseline values). | Weeks 6 and 8 of the first year (adjusted for baseline values).

SECONDARY OUTCOMES:
Quality of life (SF-36), responder rate (RQLQ score of 0.5 or more), global evaluation of treatment success, VAS (0-100 mm) overall symptom severity and nasal, eye, pharyngeal and common symptoms, safety, patients constitution, health economic analyses. | Baseline, 8 weeks and 16 weeks in the first year and baseline and week 8 in the second year

CONTACTS AND LOCATIONS:
Overall Officials: Stefan N Willich, MD, MBA, Principal Investigator — Epidemiology, and Health Economics, Charité University Medical Center, 10098 Berlin, Germany
Locations (1):
- Charité - Institute for Social Medicine, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Adam D, Grabenhenrich L, Ortiz M, Binting S, Reinhold T, Brinkhaus B. Impact of acupuncture on antihistamine use in patients suffering seasonal allergic rhinitis: secondary analysis of results from a randomised controlled trial. Acupunct Med. 2018 Jun;36(3):139-145. doi: 10.1136/acupmed-2017-011382. Epub 2018 Feb 10. PMID 29440045
- [Derived] Ortiz M, Witt CM, Binting S, Helmreich C, Hummelsberger J, Pfab F, Wullinger M, Irnich D, Linde K, Niggemann B, Willich SN, Brinkhaus B. A randomised multicentre trial of acupuncture in patients with seasonal allergic rhinitis--trial intervention including physician and treatment characteristics. BMC Complement Altern Med. 2014 Apr 6;14:128. doi: 10.1186/1472-6882-14-128. PMID 24708643
- [Derived] Reinhold T, Roll S, Willich SN, Ortiz M, Witt CM, Brinkhaus B. Cost-effectiveness for acupuncture in seasonal allergic rhinitis: economic results of the ACUSAR trial. Ann Allergy Asthma Immunol. 2013 Jul;111(1):56-63. doi: 10.1016/j.anai.2013.04.008. Epub 2013 May 3. PMID 23806461
- [Derived] Brinkhaus B, Ortiz M, Witt CM, Roll S, Linde K, Pfab F, Niggemann B, Hummelsberger J, Treszl A, Ring J, Zuberbier T, Wegscheider K, Willich SN. Acupuncture in patients with seasonal allergic rhinitis: a randomized trial. Ann Intern Med. 2013 Feb 19;158(4):225-34. doi: 10.7326/0003-4819-158-4-201302190-00002. PMID 23420231